CLINICAL TRIAL: NCT03813277
Title: Open Clinical Trial to Evaluate Safety, Tolerability, and Efficacy of Dexdor for Sedation in Paediatric Patients in Intensive Care Settings. Multi-centre Trial in Russia for Marketing Registration of Dexdor.
Brief Title: Safety, Tolerability and Efficacy of DEXDOR in Pediatric Patients in ICU
Acronym: Pedrux
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3005031
Record Dates: First submitted 2018-11-09; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: ICU Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine (Experimental): Dexmedetomidine 100microg/ml
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — infusion

SUMMARY:
Open clinical trial to evaluate safety, tolerability, and efficacy of Dexdor for sedation in paediatric patients in intensive care settings. Multi-centre trial in Russia for marketing registration of Dexdor

DETAILED DESCRIPTION:
Dexmedetomidine is in Russian currently approved for sedation only in adults; paediatric experiences in the literature are in the form of small studies and case reports.

Dexmedetomidine may be useful in paediatric patients for sedation in a variety of clinical situations. Based on literature analysis, dexmedetomidine may be potentially used in the intensive care unit in pediatric patients who require sedation, either breath spontaneously or require mechanical ventilation.

Dexmedetomidine is a newer sedative with little safety data in paediatrics, particularly for therapy lasting longer than 48 h. Additional studies in paediatric patients are warranted to further evaluate its safety and efficacy in all age ranges.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 12 to 17 years;
2. Clinical need for prolonged (>24h) light to moderate sedation in patients with spontaneous or artificial ventilation
3. Negative urine pregnancy test (for female patients);
4. Written informed consent

Exclusion Criteria:

1. Acute severe intracranial or spinal neurological disorder due to vascular causes, infection, intracranial expansion or injury; any other disorder where sedation assessment is not reliable due to any neurological conditions;
2. Uncompensated acute circulatory failure;
3. Severe hypotension or hypertension
4. Severe bradycardia or tachycardia
5. A/V-conduction block II-III;
6. Severe hepatic impairment
7. Loss of hearing or vision, or any other condition which would significantly interfere with the collection of study data;
8. Use of centrally acting alfa-2 agonists or antagonists in the period less than 5x halflife between drug discontinuation and the time of randomisation;
9. Patients who have or are expected to have treatment withdrawn or withheld due to poor prognosis
10. Patients receiving sedatives for therapeutic indications (e.g. epilepsy);
11. Patients allergic to dexmedetomidine and rescue medications
12. Hemodialysis and peritoneal dialysis;
13. Those requiring deep sedation or neuromuscular blocking agents;
14. Burn injuries and other injuries requiring regular anaesthesia or surgery;
15. History / family history of malignant hyperthermia;
16. Patients unlikely to be weaned from the ventilator during the study;
17. Patients with early-onset ventilator-associated pneumonia;
18. Any investigational drug within the preceding 30 days;
19. Any other reason which in the investigator's opinion would make it detrimental for the subject to participate in the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of Dexdor for prolonged sedation in pediatric patients | max 5 days
  Time spent in target sedation range (RASS score )
Evaluation of Dexdor efficacy for prolonged sedation in pediatric patients | max 5 days
  Proportion of patients requiring rescue medication used for inadequate sedation (rescue-medication)

SECONDARY OUTCOMES:
Wake-up/discontinuation of sedation (if applicable) | max 5 days
  Wake-up/discontinuation of sedation (if applicable)
Time to extubation. | max 5 days
  Extubation assessment (if applicable).
Time to first rescue medication | max 5 days
  Time to first rescue medication

OTHER OUTCOMES:
Safety and tolerability | max 5 days
  Clinical safety of dexdor infusion

CONTACTS AND LOCATIONS:
Overall Officials: Andershan Lekmahnov, Prof, Principal Investigator — State Federal-Funded Educational Institution of
Locations (1):
- State Federal-Funded Educational Institution of, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No